CLINICAL TRIAL: NCT00398021
Title: Predictors of Constipation in Healthy Children
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: M-2006-1168
Record Dates: First submitted 2006-11-08; First posted 2006-11-10 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2010-06

CONDITIONS: Constipation
Keywords: constipation; bowel habits
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research is to see if a questionnaire on bowel habits can help identify children who will have constipation 12 months later.

DETAILED DESCRIPTION:
Constipation in children is a common complaint, accounting for an estimated 3% of all pediatric office visits and 20% of visits to a pediatric gastroenterologist. Unfortunately, constipation can become chronic in many children even before the problem has been recognized by a parent or primary care physician. We have previously characterized the bowel habits of more than 3300 primarily middle class Caucasian children 1 to 8 years of age presenting to their primary care practitioner for a health maintenance visit. However, the validity of information concerning bowel habits of children obtained by recall is not well established. The potential benefit of this study to society will be the demonstration that a bowel habit questionnaire can predict the outcome of clinically important constipation.

ELIGIBILITY:
Inclusion Criteria:

* presenting for a health maintenance visit

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children ages 5 through 8 who present for a health maintenance visit at eleven general pediatric offices.
Sampling Method: Non-Probability Sample
Enrollment: 1430 (Estimated)
Dates: Start 2006-06; Primary Completion 2009-06 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen R Wald, MD, Principal Investigator — University of Wisconsin, Madison
Locations (11):
- United States (11):
  - Group Health Pediatrics- Capital, Madison, Wisconsin
  - UW East Pediatric Clinic, Madison, Wisconsin
  - UW East Towne Pediatrics, Madison, Wisconsin
  - Associated Physicians Pediatric Clinic, Madison, Wisconsin
  - University Station Pediatrics, Madison, Wisconsin
  - UW Pediatrics Fitchburg, Madison, Wisconsin
  - Access Community Health Centers, Madison, Wisconsin
  - UW Pediatrics-Park St., Madison, Wisconsin
  - UW West Pediatric Clinic, Madison, Wisconsin
  - UW West Towne Pediatrics, Madison, Wisconsin
  - UW Pediatrics Stoughton, Stoughton, Wisconsin

REFERENCES:
- [Background] Levine MD. Children with encopresis: A descriptive analysis. Pediatrics. 1975 Sep;56(3):412-6. PMID 1161398
- [Background] Partin JC, Hamill SK, Fischel JE, Partin JS. Painful defecation and fecal soiling in children. Pediatrics. 1992 Jun;89(6 Pt 1):1007-9. PMID 1594338
- [Background] Loening-Baucke V. Constipation in early childhood: patient characteristics, treatment, and longterm follow up. Gut. 1993 Oct;34(10):1400-4. doi: 10.1136/gut.34.10.1400. PMID 8244110
- [Background] Loening-Baucke V. Functional fecal retention with encopresis in childhood. J Pediatr Gastroenterol Nutr. 2004 Jan;38(1):79-84. doi: 10.1097/00005176-200401000-00018. PMID 14676600
- [Derived] Wald ER, Jagodzinski TD, Moyer SC, Wald A, Eickhoff JC, Edmonson MB. Validation and clinical utility of a bowel habit questionnaire in school-age children. J Pediatr Gastroenterol Nutr. 2011 Nov;53(5):520-3. doi: 10.1097/MPG.0b013e31822504fb. PMID 21617560